CLINICAL TRIAL: NCT04232488
Title: Comparison of the Distal Radial Approach Using a "Snuff Box" and the Proximal Radial Approach in Coronary Angiography and PCI
Brief Title: Distal vs Proximal Radial Approach for Coronary Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Nikola Kos, University Hospital, University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nikola1
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Coronary Disease; Vascular Diseases
Keywords: coronary disease; snuff box; radial access
MeSH Terms: conditions — Coronary Disease; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiography performed using distal radial artery (Experimental): Patients undergoing coronary angiography with or without intervention using distal radial artery ('snuff box') as a vascular access
  Interventions: Procedure: coronary angiography using distal radial artery
- Angiography performed using proximal radial artery (Active Comparator): Patients undergoing coronary angiography with or without intervention using proximal radial artery as a vascular access
  Interventions: Procedure: coronary angiography using proximal radial artery

INTERVENTIONS:
Procedure: coronary angiography using distal radial artery — Patients undergoing coronary angiography with or without percutaneous coronary intervention will be catheterised using distal radial artery ('snuff box'); color doppler will be performed after 3 months to estimate eventual occlusion of the radial artery
  Arms: Angiography performed using distal radial artery
Procedure: coronary angiography using proximal radial artery — Patients undergoing coronary angiography with or without percutaneous coronary intervention will be catheterised using proximal radial artery; color doppler will be performed after 3 months to estimate eventual occlusion of the radial artery
  Arms: Angiography performed using proximal radial artery

SUMMARY:
The distal radial approach ('snuff box' / fossa radialis) has become as valuable as the 'classical' radial approach for coronary angiography and interventions. Up to now, the success of the procedures has been described in several papers, with no difference in the complication rate and characteristics of the coronarography compared to the radial approach. It was observed that patients using distal radial access had fewer postoperative radial artery occlusions. This study will compare the characteristics of coronary angiography / percutaneous coronary intervention (duration of procedure, time to obtain the vascular arterial access, amount of contrast used, time and amount of radiation, success of procedure) and patency of radial arteries 3 months after the intervention using the distal ('snuff box') and proximal ('classic') radial approach

DETAILED DESCRIPTION:
Introduction: The distal radial approach ('snuff box' / fossa radialis) has become as valuable as the 'classical' radial approach for coronary angiography and interventions. Up to now, the success of the procedures has been described in several papers, with no difference in the complication rate and characteristics of the coronarography compared to the radial approach. It was observed that patients using distal radial access had fewer postoperative radial artery occlusions, which is particularly suitable for patients with renal disease (for preservation of the radial artery due to the potential formation of AV fistula for dialysis) and progressive coronary disease in order to preserve the radial artery for aortocoronary bypass formation. It is also potentially less likely to develop compartment syndrome and is suitable for patients with reduced forearm mobility. Since wrist immobilization during hemostatic compression is not required, the use of a distal radial approach allows for early mobilization of patients and a shorter duration of compression itself.

Aim of the study: To compare the characteristics of coronary angiography / percutaneous coronary intervention (duration of procedure, time to obtain the vascular arterial access, amount of contrast used, time and amount of radiation, success of procedure) and patency of radial arteries 3 months after the intervention using the distal ('snuff box') and proximal ('classic') radial approach Purpose of the study: to confirm the efficacy of the distal radial approach as equally effective with a lower degree of radial artery occlusion during the follow-up period Research Hypothesis: Patients using a coronary angiography / percutaneous intervention using a distal radial approach had less occlusion of the radial arteries at long-term follow-up, with no significant difference in the features of the angiography / intervention itself (duration of procedure, time to obtain the vascular access, amount of contrast used , time and amount of radiation, procedure success).

Study participants: patients undergoing coronary intervention at the Catheterization Laboratory of the Clinic for Cardiovascular Diseases at the Clinical Hospital Center "Sestre milosrdnice", Zagreb Research Methodology and Material: Standard materials and standard methods will be used to perform coronary angiography and percutaneous coronary intervention Research Plan: After signing the informed consent, the study will include 250 patients in the distal transradial approach group, and 500 patients in the proximal radial approach group (control group). The materials, as well as the procedure technique, are standardized; the characteristics of the procedure (duration of the procedure, time of obtaining the arterial access, amount of contrast used, time and amount of radiation, success of the procedure) will be observed and Doppler of the radial artery will be performed on the first following operator-specified control (usually after 3 months of the procedure) to determine the patency of the artery.

ELIGIBILITY:
Inclusion Criteria:

* signed a performed consent, older than 18 YO, clear indication for coronary angiography, palpable radial pulse

Exclusion Criteria:

* hemodynamic instability, critically ill patient, usual coronary angiography contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Occlusion of the radial artery | 3 months
  Occlusion of the radial artery used for coronary intervention diagnosed using Color Doppler